CLINICAL TRIAL: NCT03832829
Title: Evaluation of Clinical Performance and Periodontal Status of Posterior Indirect Resin Composite (Nexco) Restorations With Proximal Box Elevation Technique: A Prospective Controlled Clinical Trial up to 3 Years
Brief Title: Clinical Evaluation of Posterior Indirect Resin Composite Restorations With PBE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Collaborators: Ivoclar Vivadent AG (Industry)
Responsible Party: Principal Investigator, Funda Ozturk Bozkurt, Prof., Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 10840098-604.01.01-E.34133
Record Dates: First submitted 2019-01-29; First posted 2019-02-06 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Unsatisfactory or Defective Restoration of Tooth
MeSH Terms: interventions — Inlays

STUDY DESIGN:
Intervention Model Description: A prospective clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Indirect restorations with SR Nexco (Experimental): Large posterior defects with at least one or more cuspal coverage in molars will be restored using the materials listed (SR Nexco). Procedures will be done using local anesthesia. The procedure, starts with removal of caries or defective restorations and coronal relocation of the the margins using flowable composite with maximum thickness 1 to 1.5 mm and followed by resin composite build-up. Defined principles of morphology driven preparation technique will be followed Impression making, fabrication of indirect restoration with SR Nexco and adhesive cementation will be completed according to manufacturer's instructions.
  Interventions: Device: Indirect composite restoration

INTERVENTIONS:
Device: Indirect composite restoration — Restoration of tooth with extensive substance loss
  Other Names: Onlay and overlay restoration

SUMMARY:
Evaluation of posterior indirect resin composite restorations with proximal box elevation technique.

Restoration of large posterior defects extending below the cemento-enamel junction (CEJ) with coverage of one or more cusps represent a very common clinical situation. When restoring deep cervical margins biological and technical operative problems may occur. In order to make clinical procedures less fault-prone 'Proximal Box Elevation' (PBE) is an option that refers to application of composite resin in the deepest parts of the proximal areas in order to reposition the cervical margin supragingivally prior to cavity preparation for an indirect restoration.

This project aims to evaluate the clinical performance and periodontal status of posterior indirect composite restorations with PBE. According to study design at least 60 patients will be recruited to project and 80 restorations will be evaluated. The project will be carried out at the School of Dentistry, Istanbul Medipol University,Turkey.

DETAILED DESCRIPTION:
The rehabilitation of decayed or fractured posterior teeth using an indirect technique was introduced for large cavities with coverage of one or more cusps. Problems of biological nature and technical operative may be encountered when restoring large cavities extending below the cement-enamel junction(CEJ).

Biological problems refers to the possible violation of the 'biological width', a recommended distance of 3 mm or more between the restorative margins and the alveolar crest. The technical operative problems include difficulties in tooth preparation, impression making, adhesive cementation of the restoration, finishing and polishing in subgingival areas. In order to eliminate these difficulties Proximal Box Elevation' (PBE) was introduced that proposes application of composite resin in the deepest parts of the proximal areas in order to reposition the cervical margin supragingivally. Whether the PBE technique is the most optimal treatment option for the restoration of cavities extending below CEJ and how the proposed advantages and possible disadvantages could affect the clinical performance of the indirect restorations are the topics extensively discussed among clinicians.

According to results of in vitro studies, PBE was found to be effective in indirect resin composite bonding to deep proximal boxes in terms of marginal quality and adaptation (1).

In a retrospective clinical study, 79 indirect composite restorations were clinically examined following modified United States Public Health Service criteria. Survival rate was 91.1% and success rate was 84.8% after 5 years (2). Similarly, in another clinical study success rate of 71 indirect composite restorations was reported as 100% after 36 months (3). Nevertheless, not much scientific evidence on the influence of PBE technique on the longevity of the restorations and the periodontal health could be found in the currently available literature. Randomized controlled clinical trials with classification of baseline clinical situation and standardization of cavity preparations are necessary to evaluate the clinical performance of this technique.

This study will be carried out as a prospective study, with assessment of the restorations after three years. 80 indirect composite restorations in at least 60 patients will be included. Potential patients attending to Istanbul Medipol University Dental Clinics in Istanbul will be invited to the study. The patients meeting the inclusion criteria will be recruited. After giving their consent to take part in the study, baseline clinical situation will be classified based on technical operative and biological parameters (4).

The treatment procedure is:

Restorative process in all cases, will start with coronal relocation of the margins using flowable composite with maximum thickness 1 to 1.5 mm and followed by resin composite build-up. Defined principles of morphology driven preparation technique will be followed for standardization of cavity preparations. Impression making, fabrication of indirect restoration with SR Nexco and adhesive cementation will be completed according to manufacturer's instructions.

The control procedure is:

The restorations will be evaluated according to marginal adaptation, cavo surface marginal discoloration, approximal contact, fractures and caries associated with restorations. The periodontal status will be assessed with defined periodontal parameters. The controls will be conducted after two weeks, six months, 1year, 2 and 3 years.

ELIGIBILITY:
Inclusion Criteria:

1. Vital or endodontically treated posterior teeth with extensive substance loss
2. Caries removal or restoration replacement (i.e. amalgam, composite, glass-ionomer)
3. Large posterior defects with at least one or more cuspal coverage in molars
4. Proximal defects extending below CEJ and at least one or more cavity margin/margins located beneath the gingival tissues
5. Maximum 2 indirect restorations with SR Nexco material in each patient
6. No obvious untreated caries in the rest of the dentition, dental health problems (regularly checked by a dentist)
7. Good or moderate oral hygiene (plaque score of less than 30% in anterior region before treatment)
8. No untreated periodontal disease (only DPSI 1, 2)
9. Subjects had to be over 18 years of age, be classified according to the American Society of Anesthesiologists (ASA) as ASA I or ASA II, present with moderate to good oral hygiene, and be free of periodontal disease (probing depth and attachment levels within normal limits, no furcation involvement, and no mobility)
10. Appropriate isolation after cavity preparations
11. Subjects had to agree to keep the scheduled recall appointments for data collection and maintenance and plan to stay in the area for at least 3 years.

Exclusion Criteria:

1. Considerable horizontal and/or vertical mobility of teeth: tooth mobility index score 2 or 3 2. Considerable periodontal disease without treatment (DPSI 3-, 3+ and 4)
2. Poor endodontic prognosis
3. Pulp exposure
4. Patients who still want to bleach their teeth or bleached teeth less than 3 weeks ago
5. Extremely hypersensitive tooth
6. Excluding the teeth, without opposing natural dentition (either intact or restored with intracoronal or extracoronal fixed restorations), and with a minimum of 20 teeth
7. Substance loss due to developmental anomalies (hypoplasia, amelogenesis imperfecta etc.)
8. Subjects who presented severe wear facets and/or reported parafunctional activities such as clenching or nocturnal bruxism
9. Subjects who are pregnant or breast feeding during the duration of the study
10. Subjects who are known to be allergic to the ingredients of resin materials

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
FDI (World Dental Federation) criteria for dental restorations assessment | at 3 years
  Two independent investigators are responsible for evaluations. The primary outcome will consist in the FDI (World Dental Federation) instruments for dental restorations assessment, as it was published after consensus in 2007 and updated in 2010. This instrument is composed of three dimensions (biological, functional and esthetic), each consisting of several items that are assessed by clinical and radiographic examination according to Likert scales of 5 terms. Some items are evaluated quantitatively, others visually. The worst score of all items is retained as the overall score of the restoration, thus resulting in a single (ordinal) primary outcome.

SECONDARY OUTCOMES:
Plaque accumulation according to the Silness & Löe (1964) Plaque Index: | at 3 years
  The secondary outcome of the study relies on evaluation of periodontal status. Peridontal parameters will be scored between 0 and 3.
  0= No plaque in the gingival area.
  1. A film of plaque adhering to the free gingival margin and adjacent area of the tooth. The plaque may only be recognized by running a probe across the tooth surface.
  2. Moderate accumulation of soft deposits within the gingival pocket, on the gingival pocket, on the gingival margin and/or adjacent tooth surface, which can be seen by the naked eye.
  3. Abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.
Gingival Inflammation according to the Silness & Löe (1964) Gingival Index. | at 3 years
  0= Normal gingival.
  1. Mild inflammation-slight change in colour, slight oedema. No bleeding on probing.
  2. Moderate inflammation-redness, oedema and glazing. Bleeding on probing.
  3. Severe inflammation-marked redness and oedema. Ulceration. Tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Mutlu Özcan, DDS,PhD, Principal Investigator — University of Zurich
Locations (1):
- Istanbul Medipol University, Dental School, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hickel R, Peschke A, Tyas M, Mjor I, Bayne S, Peters M, Hiller KA, Randall R, Vanherle G, Heintze SD. FDI World Dental Federation - clinical criteria for the evaluation of direct and indirect restorations. Update and clinical examples. J Adhes Dent. 2010 Aug;12(4):259-72. doi: 10.3290/j.jad.a19262. PMID 20847997
- [Result] Juloski J, Koken S, Ferrari M. Cervical margin relocation in indirect adhesive restorations: A literature review. J Prosthodont Res. 2018 Jul;62(3):273-280. doi: 10.1016/j.jpor.2017.09.005. Epub 2017 Nov 15. PMID 29153552
- [Result] D'Arcangelo C, Zarow M, De Angelis F, Vadini M, Paolantonio M, Giannoni M, D'Amario M. Five-year retrospective clinical study of indirect composite restorations luted with a light-cured composite in posterior teeth. Clin Oral Investig. 2014;18(2):615-24. doi: 10.1007/s00784-013-1001-8. Epub 2013 May 22. PMID 23695612
- [Result] Dukic W, Dukic OL, Milardovic S, Delija B. Clinical evaluation of indirect composite restorations at baseline and 36 months after placement. Oper Dent. 2010 Mar-Apr;35(2):156-64. doi: 10.2341/09-133-C. PMID 20420058
- [Result] Veneziani M. Adhesive restorations in the posterior area with subgingival cervical margins: new classification and differentiated treatment approach. Eur J Esthet Dent. 2010 Spring;5(1):50-76. PMID 20305873
- [Derived] Aksaka N, Gozetici-Cil B, Ozcan M. Periodontal status of indirect resin composite restorations with proximal box elevation: 3-year clinical results. Clin Oral Investig. 2025 Nov 29;29(12):593. doi: 10.1007/s00784-025-06676-9. PMID 41317197